CLINICAL TRIAL: NCT04572724
Title: The Effect of Sacubitril/Valsartan on Cardiovascular Events Outcome in Maintenance Dialysis Patients With Heart Failure and Efficacy Prediction of Baseline LVEF Value：A Prospective Cohort Study
Brief Title: The Effect of Sacubitril/Valsartan on Cardiovascular Events in Dialysis Patients and Efficacy Prediction of Baseline LVEF Value
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, XUYI, Principal Investigator, Shenzhen Second People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200601054
Record Dates: First submitted 2020-09-28; First posted 2020-10-01 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Peritoneal Dialysis Complication; Hemodialysis Complication; Heart Failure
Keywords: Sacubitril/valsartan; Peritoneal dialysis; Hemodialysis; Cardiovascular Events; Efficacy Prediction
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: The participants who met the inclusion and exclusion criteria will enrolled in the trial. Subjects will be divided into two groups (1:1 matching will be achieved after a screening of propensity score) to receive one of two interventions in addition to standard HF management: Sacubitril/Valsartan group or RAS inhibitor group.
Masking Description: it is a open label cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril/Valsartan treatment group (Experimental): Sacubitril/Valsartan will be administered step by step with a titrated dose. When patients switching to Sacubitril/Valsartan from RAS inhibitor, a washout period of at least 36 hours is required to decrease the risk of angioedema.
  All subjects can have a beta-blocker, CCB, and/or alpha-blockers to control BP. Dialysis treatment: patients normally complete hemodialysis or peritoneal dialysis, need to ensure adequate dialysis requirements, no obvious overload, patients achieve dry weight after dialysis.
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet
- RAS inhibitor treatment group (Active Comparator): RAS inhibitor group allows the use of a monodose of any ACEi or ARB. All subjects can have a beta-blocker, CCB, and/or alpha-blockers to control BP. Dialysis treatment: patients normally complete hemodialysis or peritoneal dialysis, need to ensure adequate dialysis requirements, no obvious overload, patients achieve dry weight after dialysis.
  Interventions: Drug: RAS Inhibitors

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet — Sacubitril/Valsartan will start at 50mg bid, when blood pressure can be tolerable, the dose will be gradually increased to 100mg bid after taking for 2-4 weeks, and then the target dose is gradually add to the 200mg bid after another 2-4 weeks. Ensure BP>90/60mmHg, the minimum dose is 50mg bid if the patient can't tolerate higher dose but the blood pressure is stable at low dose.
  Arms: Sacubitril/Valsartan treatment group
Drug: RAS Inhibitors — RAS inhibitor group allows the use of a monodose of any ACEi or ARB. Ensure BP>90/60mmHg, the minimum dose is half dose if the patient can't tolerate monodose but the blood pressure is stable at half dose.
  Arms: RAS inhibitor treatment group

SUMMARY:
Patients with end stage renal disease (ESRD), especially after having maintenance dialysis are among the highest risk of heart failure (HF), which is the most important cause that affects survival rate and quality of life. Sacubitril/Valsartan is recommended as a first-line option for treating symptomatic chronic heart failure, especially HF with reduced ejection fraction (HFrEF). Sacubitril/Valsartan was reported the different effectiveness in HFrEF and HF with preserved ejection fraction (HFpEF), and the clinical trials' results are controversial in HFpEF patients. So far, there have been seven clinical trials (or subgroups of trials) that used sacubitril/valsartan in heart failure patients with chronic kidney disease, only one retrospective study to evaluate the improvement of cardiovascular biomarkers and LVEF in hemodialysis patients who have HFrEF. In addition, there is no article predicting the outcomes of Sacubitril/Valsartan, the inclusion criteria of LVEF value are not consistent. Investigators will perform a prospective, cohort study to evaluate the efficacy and safety of Sacubitril/Valsartan on Cardiovascular Events Outcome in Maintenance hemodialysis and peritoneal dialysis patients with Heart Failure, and use secondary analysis to find out the range of baseline LVEF Value to predict the therapeutic effects.

DETAILED DESCRIPTION:
The trial will examine the effect of Sacubitril/Valsartan on cardiovascular events in HF patients receiving maintenance hemodialysis or peritoneal dialysis. Subjects will be divided into two groups (1:1 matching will be achieved after a screening of propensity score) to receive one of two interventions in addition to standard HF management: Sacubitril/Valsartan group or RAAS inhibitor group. All subjects can have a beta-blocker, CCB, and/or alpha-blockers to control BP. Dialysis treatment: patients normally complete hemodialysis or peritoneal dialysis, need to ensure adequate dialysis requirements, no obvious overload, patients achieve dry weight after dialysis.

Participants will be treated and follow-up for at least 18 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old participants, No restrictions on gender or race
* Stable heart failure in New York Heart Association (NYHA) class II, III, or IV symptoms, presentation of typical heart failure symptoms accompanied by HF signs caused by a structural and/or functional cardiac abnormality
* Under maintenance dialysis (hemodialysis or peritoneal dialysis) for more than one year
* Patients have a plasma N-terminal pro-BNP (NT-proBNP) level ≥600 pg per milliliter, or if they had been hospitalized for heart failure within the previous 12 months, an NT-proBNP ≥400 pg per milliliter
* Patients written informed consent

Exclusion Criteria:

* Repeatedly symptomatic hypotension, systolic blood pressure of less than 90 mmHg and diastolic blood pressure of less than 60 mmHg, which cannot tolerate the RASS inhibitors therapy
* Patients who have significant fluid overload and did not reach dry weight stably
* Patients with acute myocardial infarction or implantation of intracoronary stents, coronary artery bypass grafting (CABG) and pacemaker within three months
* Patients with special type of heart disease, including cardiac amyloidosis, congential heart disease and pericardial disease
* Patients with malignant hypertension and hypertensive emergencies that can not be controlled
* Patients with significant impaired liver function
* Patients with repeatedly or server infection
* Allergic to the trial drugs
* Unacceptable side effects during receipt of RASS inhibitors
* Pregnancy
* Patients who are unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
cardiovascular events | at least 18 months
  death from any kinds of cardiovascular diseases
hospitalization for heart failure | at least 18 months
  time from the day of enroll to a first unplanned hospitalization for heart failure

SECONDARY OUTCOMES:
change rate of cardiovascular events | at least 18 months
  change rate of composite of death from cardiovascular diseases or a first unplanned hospitalization for heart failure
NT-proBNP | 12 months
  the change from baseline to 12 months in the NT-proBNP
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 1month, 6month,18 months
  the change from baseline to 1month, 6month,18 months in the clinical summary score on the Kansas City Cardiomyopathy Questionnaire (KCCQ)25 (on a scale from 0 to 100, with higher scores indicating fewer symptoms and physical limitations associated with heart failure).The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL) within a 2-week recall period. It is an important prognostic variable in cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: YI XU, Principal Investigator — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No